CLINICAL TRIAL: NCT03557437
Title: Efficacy of High Dose of Amoxicillin And Metronidazole Plus Bismuth For Helicobacter Pylori Treatment In Naive Patients : A Randomized Clinical Trial
Brief Title: High Dose of Amoxicillin and Metronidazole Plus Bismuth For Helicobacter Pylori Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjkls2018037
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori Therapy
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Therapy (Active Comparator): Esomeprazole 20mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin, Metronidazole
- Bismuth Plus Triple Therapy (Experimental): Esomeprazole 20mg bid, Bismuth Potassium Citrate 600mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin, Metronidazole; Drug: Bismuth Potassium Citrate

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Amoxicillin, Metronidazole — Antibiotics for H. pylori eradication
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Bismuth Plus Triple Therapy

SUMMARY:
Amoxicillin and metronidazole （400mg Q.D.S） based quadruple therapy had achieved a high cure rate in the rescue treatment of helicobacter pylori infection. This study aims to evaluate the efficacy and safety of the amoxicillin and metronidazole (400mg thrice a day) based triple therapy and the addition of bismuth in the naive patients with helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with no previous treatment experience

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo L, Ji Y, Yu L, Huang Y, Liang X, Graham DY, Lu H. 14-Day High-Dose Amoxicillin- and Metronidazole-Containing Triple Therapy With or Without Bismuth as First-Line Helicobacter pylori Treatment. Dig Dis Sci. 2020 Dec;65(12):3639-3646. doi: 10.1007/s10620-020-06115-7. Epub 2020 Feb 4. PMID 32020360